CLINICAL TRIAL: NCT06866249
Title: Investigation of Motor Development, Sleep Characteristics and Sensory Processing Skills of Infants With a History of Colic
Brief Title: Investigation of the Development of Infants With a History of Colic
Status: Completed | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Rabia ZORLULAR, principal investigator, Nigde Omer Halisdemir University
Other Study IDs: colic infant and development
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-03

CONDITIONS: Colic, Infantile; Motor Development; Sleep; Sensory Integration Dysfunction
Keywords: Infantile colic; developmental outcomes; motor development; sensory processing; sleep
MeSH Terms: conditions — Colic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Infantile colic: The study planned to include infants with a history of colic and their families. Evaluations will cover the demographic characteristics of the infants, sensory processing skills, motor development, and sleep patterns.
  Interventions: Behavioral: Peabody Developmental Motor Scales-2; Behavioral: Test Of Sensory Functions In Infants (Tsfı); Behavioral: Brief Infant Sleep Questionnaire
- Healthy infants: A control group consisting of healthy infants born at term with no history of colic will be established. Evaluations will include the demographic characteristics of the infants, sensory processing skills, motor development, and sleep patterns.
  Interventions: Behavioral: Peabody Developmental Motor Scales-2; Behavioral: Test Of Sensory Functions In Infants (Tsfı); Behavioral: Brief Infant Sleep Questionnaire

INTERVENTIONS:
Behavioral: Peabody Developmental Motor Scales-2 — Peabody Developmental Motor Scales | Second Edition (PDMS-2) combines in-depth assessment with training or remediation of gross and fine motor skills of children. The test is designed to identify de
Behavioral: Test Of Sensory Functions In Infants (Tsfı) — Test Of Sensory Functions In Infants (TSFI) provides objective criteria that allow you to determine whether, and to what extent, an infant has deficits in sensory functioning. Designed for use with children from 4 months to 18 months old.
Behavioral: Brief Infant Sleep Questionnaire — Infant sleep problems are among the most common problems presented to pediatricians. The extended version of the "Brief Infant Sleep Questionnaire" is a questionnaire developed by Sadeh to assess sleep problems and their causes in early childhood.

SUMMARY:
The aim of this study was to evaluate the motor development, sleep characteristics and sensory processing skills of infants with a history of colic and to compare them with their peers without a history of colic.

DETAILED DESCRIPTION:
Infantile colic (IC) is a condition characterized by incessant crying and restlessness in healthy, normally growing infants. Prolonged and intense crying in an otherwise healthy infant is a significant challenge for families. Infantile colic was first described by Wessel nearly 50 years ago. According to Wessel, episodes of crying and restlessness that last three hours a day, at least three days a week, for a minimum of three weeks are classified as infantile colic.

The long-term effects of IC include an increased risk of behavioral problems in children. A meta-analysis found that children with a history of excessive crying are more likely to develop general behavioral problems, internalizing problems (such as anxiety, depression, or withdrawal), and externalizing problems (such as aggression or disruptive behavior). Additionally, these difficulties are exacerbated by adverse family environments, including parental stress or poor maternal mental health. As these infants approach preschool age, they may struggle with sustaining attention, engaging in reciprocal play interactions, and tolerating change and separation.

The first two years of life are a critical period for supporting infant development, as brain growth and neural plasticity progress rapidly. When children reach 10-15 months of age and begin exploring their environment through walking and trial-and-error experiences, assessing sensory processing skills becomes particularly important. At this stage, children actively expand their motor repertoire, especially while developing skills such as crawling and walking. However, a review of existing studies reveals a lack of evaluations conducted during the toddler, preschool, and school-age periods. Furthermore, most studies focus primarily on behavioral problems and attention deficit hyperactivity disorder (ADHD). For this reason, 10-15-month-old infants were included in this study to assess early-stage development.

ELIGIBILITY:
Inclusion Criteria:

* Term infatns born at term
* Infants diagnosed with colic
* Post-term infants between 10-15 months

Exclusion Criteria:

* Premature infants
* Infants with congenital malformations
* Infants diagnosed with metabolic, neurological and genetic diseases
* Children whose parents do not volunteer for the study

Ages: 10 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: It was planned to include infants and families with a history of colic in the study. Children between 10-15 months of age and whose parents' consent was obtained will be included in the study.Additionally, infants and their families between 10 and 15 months of age with no history of colic will be included to compare their development.
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2025-03-12 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Peabody Developmental Motor Scales | Second Edition (PDMS-2) | 10-15 months
  Peabody Developmental Motor Scales | Second Edition (PDMS-2) in-depth assessment with training or remediation of gross and fine motor skills of children from birth through 5 years. It consists of gross motor and fine motor parts. The Gross motor section includes 151 items from 4 subtests: reflexes, stasis, locomotion, and object manipulation. The fine motor section consists of 2 subtests and 98 items: comprehension and visual-motor integration. The total motor part is the sum of the items in the gross and fine 25 motor parts. Items are scored with 0, 1, and 2 points. When the child performs the item according to the specified item criteria, 2 points are given. One point is awarded when the behavior occurs, but the criteria for successful performance are not fully met. A score of 0 is given when the child is unable to try the item or does not reveal any skills when he tries it. Results are expressed as raw, standard, or total motor scores.
Test of Sensory Functıons ın Infants | 10-15 months
  This test helps you identify infants with sensory integrative dysfunction-including those at risk for developing learning disabilities as they grow older. All subtests consist of a total of 24 items. In the tactile deep pressure response section, it is scored as 0: reverse response, 1: mild defensive response, and 2: integrated response. In the adaptive motor response section, it is scored as 0: no response, 1: disorganized, 2: partial, 3: organized. In the visual-tactile integration section, it is scored as 0: hyperactive, 1: hyporeactive, and 2: normal. The oculomotor test section is scored as 0: no response or poorly integrated, 1: well integrated. Response to vestibular stimulation is scored as 0: adverse response, 1: mild defensive response, and 2: integrated response. The total score ranges from 0 to 49. In 10-12-month-old babies, 44-49 points indicate good sensory function, 41-43 points indicate risky status, 0-40 points sensory processing problem.
Brief Infant Sleep Questionnaire | 10-15 months
  The Brief Infant Sleep Questionnaire will be used to assess sleep. Infant sleep problems are among the most common problems presented to pediatricians. The extended version of the "Brief Infant Sleep Questionnaire" is a questionnaire developed by Sadeh to assess sleep problems and their causes in early childhood. This questionnaire has been translated into Turkish and assessed sleep environment and sleep problems in infants. It consists of 33 items, is based on parental reports of infant or toddler sleep patterns and is used to validate the data. It is associated with daily records and parental sleep reports. Its sensitivity in documenting developmental sleep trends is well established

CONTACTS AND LOCATIONS:
Overall Officials: Rabia ZORLULAR, Principal Investigator — Nigde Omer Halisdemir University
Locations (2):
- Turkey (Türkiye) (2):
  - Gazi University, Ankara
  - Nigde Omer Halisdemir University, Niğde

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeGangi, G.A. and S.I. Greenspan, The development of sensory functions in infants. Physical & Occupational Therapy in Pediatrics, 1989. 8(4): p. 21-33
- [Background] Boran, P., et al., Translation into Turkish of the expanded version of the "Brief Infant Sleep Questionnaire" and its application to infants. Marmara Medical Journal, 2014. 27(3): p. 178-183.
- [Background] Folio, M.R., Peabody developmental motor scales. DLM Teaching Resources, 1983.
- [Background] Canivet C, Jakobsson I, Hagander B. Infantile colic. Follow-up at four years of age: still more "emotional". Acta Paediatr. 2000 Jan;89(1):13-7. doi: 10.1080/080352500750028988. PMID 10677050